CLINICAL TRIAL: NCT00320450
Title: A Randomised, Parallel Group, Placebo-controlled, Double Blind Study to Assess the Safety and Tolerability of SB-681323 at 7.5mg Daily Dose for 28 Days and Its Effect on the Levels of Serum C-reactive Protein (CRP) in Subjects With Rheumatoid Arthritis (RA)
Brief Title: SB-681323 In Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RA1100849
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2012-05

CONDITIONS: Arthritis, Rheumatoid
Keywords: SB-681323; CRP; Rheumatoid Arthritis SB-681323 CRP RA; Rheumatoid Arthritis; RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — dilmapimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB-681323

SUMMARY:
The purpose of this research is to find out how effective and safe SB-681323 will be in the treatment of RA when it is added to standard anti-rheumatic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Females cannot be pregnant or lactating.
* Must use defined contraceptive methods if of child-bearing potential.
* BMI range: 18.5-35.0 kg/m2.
* Diagnosis of RA (rheumatoid arthritis) according to revised 1987 American College of Rheumatology (ACR) criteria.
* If other RA-medication is used: Disease-Modifying Anti-Rheumatic Drug (DMARDS) must be stable for at least 8 weeks before first trial visit.
* If other oral anti-RA therapies are used, these must have been stable at least 4 weeks before first trial visit.
* If Methotrexate medication is used as RA-therapy, Folate supplement must be taken with stable red cell folate levels.
* Must give informed consent.
* Must abstain from alcohol during the trial participation.

Exclusion Criteria:

* Non-responder on biological RA treatment.
* Has a positive alcohol screen.
* Any history of liver disease.
* Positive Hepatitis B surface antigen or Hepatitis C antibody result within 3 months of screening.
* Have any significant disease that places the subject at unacceptable risk as a participant in this trial.
* Acute infection.
* History of active tuberculosis.
* History of repeated or chronic infection.
* History of malignancy.
* History of HIV or other immunosuppressive diseases.
* Participated in a clinical trial within the last 3 months for non-biological therapies and 6 months for biological therapies.
* Uncontrolled diabetes or psoriasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2005-11; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Serum levels of CRP at the end of study (after 28 days of treatment) following repeat dosing with SB-681323 (7.5mg/day) compared with placebo. | 28 Days

SECONDARY OUTCOMES:
Serum levels of CRP at other available timepoints. The following secondary endpoints will be analysed at all available timepoints: Clinical Symptoms, Safety and Biomarkers, Health Outcome. | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (39):
- GSK Investigational Site, Hvidovre, Denmark
- Germany (8):
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hofheim, Hesse
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
- GSK Investigational Site, Shatin, Hong Kong
- Italy (5):
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Benevento, Campania
  - GSK Investigational Site, Telese Terme (BN), Campania
  - GSK Investigational Site, Jesi (AN), The Marches
  - GSK Investigational Site, Pisa, Tuscany
- Norway (6):
  - GSK Investigational Site, Drammen
  - GSK Investigational Site, Lillehammer
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Sarpsborg
  - GSK Investigational Site, Stavanger
  - GSK Investigational Site, Tønsberg
- Poland (3):
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Spain (8):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Baracaldo/Vizcaya
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Mérida
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- Sweden (2):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Luleå
- United Kingdom (5):
  - GSK Investigational Site, Wigan, Lancashire
  - GSK Investigational Site, Metropolitan Borough of Wirral, Merseyside
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, London
  - GSK Investigational Site, Sheffield